CLINICAL TRIAL: NCT02735603
Title: A Randomized, Double-Blind, Placebo- and Moxifloxacin Positive-Controlled (Open-Label), Cross-Over Study to Evaluate the Potential Effect of Naltrexone and Bupropion Extended-Release Combination on Cardiac Repolarization in Healthy Subjects
Brief Title: Study to Evaluate the Effect of Naltrexone and Bupropion Extended-Release Combination on Cardiac Repolarization in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orexigen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: NaltrexBuprop-1001; U1111-1171-3290 (Registry Identifier: WHO)
Record Dates: First submitted 2016-04-05; First posted 2016-04-12 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Heart Repolarization
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Nalterxone/Bupropion + Placebo + Moxifloxacin (Experimental): Naltrexone hydrochloride (HCl) 8 milligram (mg)/bupropion HCl 90 mg (NB) placebo-matching 2 tablets, orally, once in the morning on Day -1, NB, 1 extended-release tablet, orally, twice daily and NB placebo-matching 1 tablet, orally, twice daily from Days 1 to 3, NB, 2 extended-release tablets, orally, twice daily from Days 4 to 10 and once in the morning on Day 11 in treatment period 1, followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10, and once in the morning on Day 11 in treatment period 2, followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10, moxifloxacin 400 mg, tablet, orally, once in the morning on Day 11 in treatment period 3.
  Interventions: Drug: Naltrexone HCl/bupropion HCl; Other: Placebo; Drug: Moxifloxacin
- Placebo + Moxifloxacin + Naltrexone/Bupropion (Experimental): NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10 and once in the morning on Day 11 in treatment period 1, followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10, moxifloxacin 400 mg, tablet, orally, once in the morning on Day 11 in treatment period 2, followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, NB, 1 extended-release tablet, orally, twice daily and NB placebo-matching 1 tablet, orally, twice daily from Days 1 to 3, NB, 2 extended-release tablets, orally, twice daily from Days 4 to 10 and once in the morning on Day 11 in treatment period 3.
  Interventions: Drug: Naltrexone HCl/bupropion HCl; Other: Placebo; Drug: Moxifloxacin
- Moxifloxacin + Naltrexone/Bupropion + Placebo (Experimental): NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10, moxifloxacin 400 mg, tablet, orally, once in the morning on Day 11 in treatment period 1, followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, NB, 1 extended-release tablet, orally, twice daily and NB placebo-matching 1 tablet, orally, twice daily from Days 1 to 3, NB, 2 extended-release tablets, orally, twice daily from Day 4 to 10, and once in the morning on Day 11 in treatment period 2, followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10 and once in the morning on Day 11 in the treatment period 3.
  Interventions: Drug: Naltrexone HCl/bupropion HCl; Other: Placebo; Drug: Moxifloxacin
- Naltrexone/Bupropion + Moxifloxacin + Placebo (Experimental): NB placebo-matching 2 tablets, orally, once in the morning on Day -1, NB, 1 extended-release tablet, orally, twice daily and NB placebo-matching 1 tablet, orally, twice daily from Days 1 to 3, NB, 2 extended-release tablets, orally, twice daily from Days 4 to 10 and once in the morning on Day 11 in treatment period 1, followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10, moxifloxacin 400 mg, tablet, orally, once in the morning on Day 11 in treatment period 2 followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10 and once in the morning on Day 11 in treatment period 3.
  Interventions: Drug: Naltrexone HCl/bupropion HCl; Other: Placebo; Drug: Moxifloxacin
- Placebo + Naltrexone/Bupropion + Moxifloxacin (Experimental): NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10 and once in the morning on Day 11 in treatment period 1, followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, NB, 1 extended-release tablet, orally, twice daily and NB placebo-matching 1 tablet, orally, twice daily from Days 1 to 3, NB, 2 extended-release tablets, orally, twice daily from Days 4 to 10 and once in the morning on Day 11 in treatment period 2 followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10, moxifloxacin 400 mg, tablet, orally, once in the morning on Day 11 in treatment period 3.
  Interventions: Drug: Naltrexone HCl/bupropion HCl; Other: Placebo; Drug: Moxifloxacin
- Moxifloxacin + Placebo + Naltrexone/Bupropion (Experimental): NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10, moxifloxacin 400 mg, tablet, orally, once in the morning on Day 11 in treatment period 1 followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, twice daily from Days 1 to 10 and once in the morning on Day 11 in treatment period 2 followed by 14 days washout period, followed by NB placebo-matching 2 tablets, orally, once in the morning on Day -1, NB, 1 extended-release tablet, orally, twice daily and NB placebo-matching 1 tablet, orally, twice daily from Days 1 to 3, NB, 2 extended-release tablets, orally, twice daily from Days 4 to 10 and once in the morning on Day 11 in treatment period 3.
  Interventions: Drug: Naltrexone HCl/bupropion HCl; Other: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Naltrexone HCl/bupropion HCl — Naltrexone HCl/bupropion HCl extended-release tablet.
Other: Placebo — Naltrexone/bupropion placebo-matching tablets.
Drug: Moxifloxacin — Moxifloxacin tablet.

SUMMARY:
The purpose of this study is to evaluate the potential effect of naltrexone and bupropion extended-release combination on cardiac repolarization in healthy participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called naltrexone HCl/bupropion HCl (NB). NB is approved by the U.S. Food and Drug Administration (FDA) in addition to a reduced-calorie diet and increased physical activity for chronic weight management in adults who are obese or who are overweight and have at least one additional weight-related condition such as high blood pressure, diabetes or high cholesterol. This study is conducted to determine the potential effect of NB relative to placebo on cardiac repolarization.

The study will enroll approximately 84 participants. Participants will be randomly assigned (by chance, like flipping a coin) to 1 of 6 treatment sequences, which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Naltrexone/Bupropion + Placebo + Moxifloxacin
* Placebo + Moxifloxacin + Naltrexone/Bupropion
* Moxifloxacin + Naltrexone/Bupropion + Placebo
* Naltrexone/Bupropion + Moxifloxacin + Placebo
* Placebo + Naltrexone/Bupropion + Moxifloxacin
* Moxifloxacin + Placebo + Naltrexone/Bupropion

This study is consisted of 3 periods separated by a washout period (Days 11 through 25). Participants will be admitted to the clinic on Day -2 (Check-in) of each study period and will remain confined to the clinic until the morning of Day 12 of each study period. On Day -1 and Day 11 of each period, participants will undergo 24 hour Holter recordings using an ambulatory electrocardiograph recorder.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 96 days.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male or female.
2. Is aged 18 to 55 years, inclusive, at signing of informed consent and first dose of study drug.
3. Weighs at least 50 kilogram (kg) and has a body mass index (BMI) of 18.0 to 35.0 kilogram per square meter (kg/m^2), inclusive, at screening.

Exclusion Criteria:

1. Has known hypersensitivity to moxifloxacin or other quinolone antibiotics or any component of the formulation of naltrexone/bupropion.
2. Has a history of seizure of any etiology, or of predisposition to seizures.
3. Has a history of significant cardiac disease.
4. Has a history of bulimia.
5. Has a history of anorexia nervosa.
6. Has a hemoglobin concentration less than (<) 12 gram per deciliter (g/dL) at screening or check-in (day -2) of period 1.
7. Has resting heart rate outside the normal range of 45 to 100 beats per minute at screening or check-in (day -2) of period 1.
8. Has orthostatic blood pressure greater than or equal to (>=) 25 millimeters of mercury (mm Hg) at screening or check-in (day -2) of period 1.
9. Has sustained supine systolic blood pressure >=140 mm Hg or <=90 mm Hg or a diastolic blood pressure >=90 mm Hg or <=50 mm Hg at screening or check-in (day -2) of period 1.
10. Has abnormal screening or check-in (day -2) of period 1 ECG indicating a second- or third-degree atrioventricular block, or 1 or more of the following: PR >220 msec, QRS >120 msec, and QTcF >450 msec, or any rhythm other than sinus rhythm that is interpreted by the investigator to be clinically significant or could interfere with an accurate measurement of the QT interval.
11. Has family history of long QT syndrome.
12. Had extensive exercising in normal life, for example, marathon running, triathlon, physical sports at a contest level.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The time-matched change from Baseline in QT interval with Fridericia correction method (QTcF) | Time matched Baseline and Day 11 within 30 minutes predose and up to 23.5 hours postdose
  QT and RR intervals will be recorded using ECG machines. Fridericia correction method is calculated by dividing QT interval by the cube root of the RR interval: QTcF = QT/RR^1/3.

SECONDARY OUTCOMES:
Time-Matched Change From Baseline in QT Interval With Bazett Correction Method (QTcB) at Day 11 | Time matched baseline and at multiple time-points (up to 23.5 hours) postdose on Day 11
  QT and RR intervals will be recorded using ECG machines. QTcB will be calculated by dividing QT interval by the square root of the RR interval: QTcB = QT/RR^1/2.
Time-Matched Change From Baseline in QT Interval With Individual Correction Method (QTcI) at Day 11 | Time matched baseline and at multiple time-points (up to 23.5 hours) postdose on Day 11
  QT and RR intervals will be recorded using ECG machines. QTcI will be calculated as QT/RR^beta, where the value of beta will be calculated using linear regression modeling for each subject on all baseline QT - RR interval pairs.
Time-Matched Change From Baseline in Uncorrected QT at Day 11 | Time matched baseline and at multiple time-points (up to 23.5 hours) postdose on Day 11
Time-Matched Increases From Baseline in QTcF, QTcB, QTcI, and QT > 30 msec and > 60 msec at Day 11 | Baseline and Day 11
  QTcF will be calculated by dividing QT interval by the cube root of the RR interval: QTcF= QT/RR^1/3. QTcB will be calculated by dividing QT interval by the square root of the RR interval: QTcB = QT/RR^1/2. QTcI will be calculated as as QT/RR^beta, where the value of beta will be calculated using linear regression modeling for each subject on all baseline QT - RR interval pairs
QTcF, QTcB, QTcI, and QT intervals >450 msec, >480 msec or >500 msec at Day 11 | Day 11
  QTcF will be calculated by dividing QT interval by the cube root of the RR interval: QTcF= QT/RR^1/3. QTcB will be calculated by dividing QT interval by the square root of the RR interval: QTcB = QT/RR^1/2. QTcI will be calculated as QT/RR^beta., where the value of beta will be calculated using linear regression modeling for each subject on all baseline QT - RR interval pairs.
T-U wave complex morphology on Day 11 | Day 11
Cmax- Maximum Observed Plasma Concentration for Naltrexone, Bupropion, and their Metabolites | Day 11: predose and at multiple time points (up to 23.5 hours) postdose
Tmax- Time to Reach the Maximum Plasma Concentration (Cmax) for Naltrexone, Bupropion, and their Metabolites | Day 11: predose and at multiple time points (up to 23.5 hours) postdose
9. Percentage of Participants Reporting at least one Treatment-Emergent Adverse Event (TEAE) | Baseline up to 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Austin, Texas, United States